CLINICAL TRIAL: NCT03240146
Title: Pulsed Shortwave Therapy (PSWT) Treatment for Chronic Musculoskeletal Low Back Pain
Brief Title: Pulsed Shortwave Therapy Treatment for Chronic Musculoskeletal Low Back Pain
Acronym: PSWT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioElectronics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SAIRB-17-0057
Record Dates: First submitted 2017-08-02; First posted 2017-08-04 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Devices will be coded, the placebo device is Identical to the active device in all ways except emitting the electromagnetic field. The energy emitted causes no sensation so can not be unmasked by user.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Study Group (Active Comparator): Subjects in this group will receive an active pulsed shortwave therapy device.
  Interventions: Device: Pulsed Shortwave Therapy
- Control Group (Placebo Comparator): Subjects in this group will receive a placebo pulsed shortwave device that it does not emit energy.
  Interventions: Device: Pulsed Shortwave Therapy

INTERVENTIONS:
Device: Pulsed Shortwave Therapy — Pulsed Shortwave Therapy device

SUMMARY:
The ActiPatch is a cutaneous device which is CE marked approved for relief of pain and has FDA clearance as an over the counter device for the adjunctive treatment of osteoarthritis of the knee and plantar fasciitis. It is taped over the affected area and stimulation at a high frequency is reported to alleviate pain with no sensation. By randomising patients between application of an active device or a dummy device and assessment of disability and pain scores at four weeks the efficacy or otherwise can be established. Chronic low back pain is a major health problem and if effective this has major economic implications as the device is cheap and safe.

DETAILED DESCRIPTION:
Chronic low back pain is a major public heath challenge for a number of reasons including prevalence, seriousness, vulnerable populations, the utility of population health strategies, and the importance of prevention at both the population and individual levels. Its incidence and prevalence are increasing with an aging population and the rise in obesity. When considering the location of chronic pain and its aetiology, back pain was the most common location with arthritis/osteoarthritis being the most common cause. Chronic low back back pain is costly to nations-not just in terms of health care expenditures and disability compensation but also in terms of lost school days, lost productivity and employment, reduced incomes, and lost potential and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial.
* In the Investigator's opinion, is able and willing to comply with all trial requirements.
* Male or female ages 18 or above with stable chronic lower back pain
* Females of childbearing must be on birth control or practice abstinence during the study period

  o Women of childbearing age will be screened with a urine pregnancy test. Women of childbearing potential are defined as any female who has experienced menarche and who is not permanently sterile or postmenopausal. Postmenopausal is defined as 12 consecutive months with no menses without an alternative medical cause.
* ≥3 months duration of chronic low back pain
* a current VAS pain rating ≥5/10
* no radiating pain below the knee
* Most of the pain in the body is present in the lower back or buttock, NOT in the lower extremities, as determined during screening by the principal investigator. The investigator will verbally ask the participant if most of the pain being experienced is in the lower back/buttock area, and rely on the response for inclusion into the study.
* able to complete and tolerate treatment for the study period.

Exclusion Criteria:

* Female participant who is pregnant.
* Significant renal or hepatic impairment confirmed by medical history.
* Prior home use of pulsed shortwave therapy.
* Prior history of spinal fusion or failed spinal surgery syndrome.
* Laminectomy, laminotomy or discectomy within 12 months of enrollment.
* Diagnostic or interventional injections or any low back surgeries not mentioned above, including radiofrequency neuroablation within 6 months of enrollment.
* The addition of strong opiates (hydrocodone, oxycodone, morphine), pregabalin and gabapentin to the treatment regime during the course of the trial
* Current implanted cardiac demand pacemakers, defibrillators, cardiac pumps, spinal stimulators or other implanted electronic devices.
* Patients using personal home based electrical stimulation devices are excluded
* Patients with other concomitant illnesses (e.g., malignancy, osteoporosis) which, in the opinion of the investigator, would preclude successful patient participation will also be excluded
* Active psychiatric disorders will be excluded (e.g. use of antipsychotic medication, bipolar disorder, schizophrenia).
* Patients diagnosed with history of significant mood disorder will be excluded (e.g., depression or anxiety with adequate control would be acceptable).
* Scheduled elective surgery or other procedures requiring general anaesthesia during the trial.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Participants who have participated in another research trial involving an investigational product in the past 12 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index | 4 weeks
  Quality of life measure for chronic lower back pain

SECONDARY OUTCOMES:
Visual Analogue Pain score | 4 weeks
  assessment of pain being experienced
The Pain and Sleep Questionnaire three-item index | 4 weeks
  Assessment of the impact of pain on the subjects sleep
Analgesic Medication use | 4 weeks
  Quantify the use of analgesic medications

CONTACTS AND LOCATIONS:
Overall Officials: Chandra Koneru, MD, Principal Investigator — North Alabama Primary Care; Sree Koneru, Ph.D, Study Director — BioElectronics Corporation; Ian Rawe, Ph.D., Study Chair — BioElectronics Corporation
Locations (1):
- North Alabama Primary Care, Athens, Alabama, United States

IPD SHARING:
Plan to Share IPD: No